CLINICAL TRIAL: NCT06927791
Title: MAchine Learning to Boost the Early Diagnosis of Acute Cardiovascular Conditions
Acronym: MALBEC
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University of Basel (Other)
Responsible Party: Sponsor
Other Study IDs: kt25boeddinghaus
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Acute Cardiovascular Disease; ST-segment Elevation Myocardial Infarction (STEMI); NSTEMI - Non-ST Segment Elevation MI
Keywords: Machine Learning; Clinical Decision Support Tool; Cardiac Biomarkers; Deep Transfer Learning (DTL); Artificial Intelligence; Acute cardiovascular conditions
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with acute chest pain and/or acute dyspnoea: Patients with acute chest pain and/or acute dyspnoea
  Interventions: Other: Machine learning based development of a diagnostic tool for acute cardiovascular disease

INTERVENTIONS:
Other: Machine learning based development of a diagnostic tool for acute cardiovascular disease — MALBEC will be delivered through five integrated work packages (WP) encompassing: (0) platform development and implementation, (1) data pooling, (2) model development, (3) performance comparison, (4) performance validation, and (5) platform plugin

SUMMARY:
The research project aims to develop clinical decision support tools integrating established diagnostic variables and machine learning (ML) models for rapid diagnosis of acute life-threatening cardiovascular conditions in emergency department (ED) patients with chest pain or dyspnea with the ultimate goal of Improved diagnostic accuracy, faster patient management, and reduced medical errors.

DETAILED DESCRIPTION:
Current State of Research in the Field

Acute cardiovascular disease (ACVD) is the leading cause of death in Switzerland and Europe, responsible for 29% of deaths in Switzerland and 36% across Europe. The increasing prevalence of ACVD, including acute myocardial infarction (AMI), acute heart failure (AHF), pulmonary embolism (PE), and acute aortic syndromes (AAS), places a significant burden on healthcare systems. Diagnosing these conditions in emergency departments (EDs) is challenging due to overlapping symptoms and the need for rapid, accurate decision-making.

The introduction of cardiovascular biomarkers, including high-sensitivity cardiac troponin, B-type natriuretic peptide, and D-dimer has revolutionized early diagnosis. These biomarkers, alongside clinical assessments and electrocardiograms (ECGs), are now essential diagnostic tools. However, current diagnostic algorithms have still tremendous limitations.

Recent advances in machine learning (ML) and deep learning (DL) offer opportunities to improve diagnosis. ML-based ECG interpretation and deep transferable learning (DTL) techniques could enhance diagnostic accuracy by integrating complex ECG and biomarker data. AutoML approaches can further refine these models, reducing human error and improving clinical workflows.

The research team has conducted multiple large-scale studies leading to significant advancements in cardiovascular biomarker research and precision medicine. Their contributions include:

* Validation of the MI3 model, which uses ML to improve NSTEMI
* Introduction of the BASEL ECG Score, a quantitative tool that enhances NSTEMI diagnosis.
* Validation of CoDE-ACS, an ML-based clinical decision support-tool that predicts the probability of NSTEMI more effectively than standard cardiac troponin thresholds.

The team is now focussing on integrating ECG data with biomarkers using AI/ML to enhance accuracy and automate decision-making. Collaboration with international experts has enabled the successful application of neural networks to ECG interpretation. The next steps include:

* Refining ML-based ECG interpretation to incorporate non-additive effects.
* Expanding ML models to include multiple cardiovascular conditions beyond AMI.
* Integrating these AI-driven tools into clinical workflows and electronic health records.

This research aims to revolutionise cardiovascular diagnostics by leveraging AI and ML for more precise, faster, and clinically relevant decision-making.

Objectives:

1. Develop and implement a clinical decision support tool that visualizes key diagnostic data.
2. Train and validate ML models to diagnose acute cardiovascular diseases (ACVD).
3. Compare ML model performance with existing diagnostic algorithms.
4. Validate ML models in large international clinical trials.
5. Integrate ML models into the electronic patient record at the University Hospital Basel.

ELIGIBILITY:
Inclusion Criteria:

• Acute cardiovascular disease (ACVD)

Exclusion Criteria

* age < 18 years old
* patients presenting in cardiogenic shock
* chronic terminal kidney failure requiring dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dataset of about 200'000 extensively characterized patients enrolled in randomized controlled trials and observational studies are used
Sampling Method: Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Developing a clinical decision support tool | During whole study duration of 3 years
  Developing and implementing a clinical decision support tool that integrates and visualizes results of established diagnostic variables in a dashboard
Validate machine learning (ML) models | During whole study duration of 3 years
  Derive and validate ML models that integrate cardiac biomarkers with key clinical information and the digital 12-lead ECG to rapidly inform the diagnostic probability for six acute life-threatening cardiovascular conditions in patients presenting with acute chest pain and/or acute dyspnoea to the Emergency Department

CONTACTS AND LOCATIONS:
Overall Officials: Christian Müller, Prof. Dr. med., Study Director — University Hospital, Basel, Switzerland; Jasper Boeddinghaus, PD Dr. med., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No